CLINICAL TRIAL: NCT03456518
Title: Pattern of Acute on Chronic Liver Failure in Patient With HCV Related Chronic Liver Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Khaled, resident doctor, Assiut University
Other Study IDs: POACLIFWHCV LC
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The concept of acute-on-chronic liver failure (ACLF) was introduced by Jalan and Williams in 2002 to describe the acute deterioration in liver function over 2 to 4 weeks in a patient with well-compensated cirrhosis associated with a precipitating event (hepatotoxic: superimposed hepatitis viral infection, drug-induced liver injury, hepatotoxins, or excessive alcohol consumption; extra hepatic: variceal bleeding or sepsis), leading to severe deterioration in clinical status with jaundice and hepatic encephalopathy and/or HRS. Following this concept, several proposals for the diagnostic criteria of ACLF have been suggested.

DETAILED DESCRIPTION:
There may be regional differences in etiology, pathogenesis, and natural course of ACLF, which may in turn influence the overall outcome of this syndrome. So, proper diagnosis of ACLF and its precipitating factors in our locality enable us for proper management of these cases and dealing with these precipitating factors to be avoided later on in patients with liver cirrhosis

Aim of the work:

To identify the pattern of acute on chronic liver cell failure (ACLF) within 28 days including prevalence, percipitating factors, and outcome.

Patients and methods

Type of the study: Prospective hospital based study

Site of the study: Tropical Medicine and Gastroenterology Department, Al-Rajhi University Hospital, Assiut University Hospitals, Assiut, Egypt. Written consent will be obtained from all the participants or their relatives before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with HCV related CLD based on clinical, biochemical and imaging evidence., with or without prior decompensation.
* Patients diagnosed to have ACLIF at any grade (1-3)

Exclusion Criteria:

* Acute liver failure without evidence of chronic liver disease.
* Other etiology of chronic liver disease
* Patients diagnosed with no ACLIF No ACLF
* This category includes patients who either:

  * Do not have any organ failure
  * Have a single organ failure that does not involve the kidney with a serum creatinine level of <1.5 mg per dl and no hepatic encephalopathy
  * Have a single brain failure with a serum creatinine level of <1.5 mg per dl
* Patients refuse to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: CLD patients with HCV related etiology who will admitted to our hospital with picture of acute decompensation and deterioiration of pre-existing liver condition (defined by the development of ascites, encephalopathy, gastrointestinal haemorrhage and/or bacterial infection) associated with either a single organ failure (single renal failure or other single non-renal organ failure if associated with renal and/or brain dysfunction) or multiple organ failures) to meet the criteria of EASL-CLIF definition .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
pattern of acute on chronic liver cell failure | march 2018 to march 2019
  evaluation of cases with acute on chronic liver cell failure as number of cases diagnosed with ACLF in this period , the precipitating factor of the condition , the fate of the patient (improving or deterioration or death ) in the 28 days following diagnosis .

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Medhat, Study Director — Al-Arajhy Liver Hospital, Assiut University
Locations (2):
- Egypt (2):
  - Al-Rajhi Liver Hospital, Assiut University, Asyut
  - Al-Rajhi liver hospital ,Assiut university, Asyut

REFERENCES:
- [Background] Gines P, Quintero E, Arroyo V, Teres J, Bruguera M, Rimola A, Caballeria J, Rodes J, Rozman C. Compensated cirrhosis: natural history and prognostic factors. Hepatology. 1987 Jan-Feb;7(1):122-8. doi: 10.1002/hep.1840070124. PMID 3804191